CLINICAL TRIAL: NCT02686762
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled Trial of Emricasan (IDN-6556-12), an Oral Caspase Inhibitor, in Subjects With Non-alcoholic Steatohepatitis (NASH) Fibrosis
Brief Title: Emricasan, a Caspase Inhibitor, for Evaluation in Subjects With Non-Alcoholic Steatohepatitis (NASH) Fibrosis
Acronym: ENCORE-NF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDN-6556-12
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Non-alcoholic Steatohepatitis; Fibrosis; Liver Diseases
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Liver Diseases | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Emricasan (5 mg) (Active Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Fibrosis will be administered orally with emricasan (5 mg) twice a day.
  Interventions: Drug: Emricasan (5 mg)
- Emricasan (50 mg) (Active Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Fibrosis will be administered orally with emricasan (50 mg) twice a day.
  Interventions: Drug: Emricasan (50 mg)
- Matching Placebo (Placebo Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Fibrosis will be administered orally with a matching placebo twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emricasan (5 mg) — Subjects with Non-alcoholic Steatohepatitis (NASH) Fibrosis will be administered orally with emricasan (5 mg) twice a day.
  Other Names: IDN-6556
  Arms: Emricasan (5 mg)
Drug: Emricasan (50 mg) — Subjects with Non-alcoholic Steatohepatitis (NASH) Fibrosis will be administered orally with emricasan (50 mg) twice a day.
  Other Names: IDN-6556
  Arms: Emricasan (50 mg)
Drug: Placebo — Subjects with Non-alcoholic Steatohepatitis (NASH) Fibrosis will be administered orally with a matching placebo twice a day.
  Arms: Matching Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled trial involving subjects with a diagnosis of "definite NASH" with fibrosis (excluding cirrhosis) as determined by the central histopathologist. Upon successful screening, subjects will be randomized to receive either emricasan 50 mg BID or emricasan 5 mg BID or matching placebo BID.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older, able to provide written informed consent, and able to understand and willing to comply with the requirements of the study
2. Histological evidence of definite NASH based on NASH CLinical Research Network (CRN) criteria, as confirmed by the central histopathologist, on a liver biopsy obtained no more than 6 months prior to Day 1
3. NAFLD Activity Score (NAS) of 4 or greater with a score of at least 1 in each component of the NAS (steatosis scored 0-3, lobular inflammation scored 0-3, ballooning scored 0-2)
4. Fibrosis stage 1 (limited to 20% of subjects), stage 2, or stage 3 using the NASH CRN Histologic Scoring System

   a. Subjects with fibrosis stage 1 must also have diabetes mellitus or metabolic syndrome
5. Willingness to utilize effective contraception (for both males and females of childbearing potential) from Screening to 4 weeks after the last dose of study drug
6. If on vitamin E or pioglitazone, subjects must have been on a stable dose for at least 3 months prior to the biopsy (whether historical or qualifying biopsy)

Exclusion Criteria:

1. Current or history of significant alcohol consumption, defined as more than 20 g/day for females and more than 30 g/day in males on average, or inability to reliably quantify alcohol consumption based on investigator's judgement
2. Use of the following drugs (which may have potential hepatotoxic effects) within 6 months prior to Day 1: amiodarone, methotrexate, tamoxifen, valproic acid, estrogens at doses greater than those used for hormone replacement or contraception, anabolic steroids, or systemic glucocorticoids for more than 4 weeks at doses greater than replacement doses
3. Uncontrolled diabetes (HbA1c ≥9%) within 60 days prior to Day 1
4. Presence of cirrhosis on liver biopsy (fibrosis stage 4 based on the central histopathologist reading)
5. Hepatitis and fibrosis more likely related to etiologies other than NASH such as:

   1. alcoholic steatohepatitis
   2. autoimmune hepatitis
   3. hepatitis B virus (HBV) infection
   4. hepatitis C virus (HCV) infection
   5. primary biliary cirrhosis
   6. primary sclerosing cholangitis
   7. Wilson's disease
   8. alpha-1-antitrypsin deficiency
   9. hemochromatosis or iron overload
   10. drug-induced liver disease
   11. other biliary liver disease
6. ALT or AST >5 times upper limit of normal (ULN) or total bilirubin >1.5 times ULN during screening (unless subject has elevated total bilirubin due to Gilbert's as documented in the medical records)
7. Alpha-fetoprotein >200 ng/mL
8. Hemoglobin <10 g/dL
9. White blood cell count <2.0 x 10^3/mm3
10. Estimated creatinine clearance <30 mL/min
11. Current use of the following medications that are considered significant inhibitors of OATP1B1 and OATP1B3 transporters: atazanavir, cyclosporine, eltrombopag, gemfibrozil, indinavir, lopinavir, ritonavir, rifampin, saquinavir, simeprevir, telaprevir, tipranovir, or some combination of these medications
12. Symptoms of biliary colic, e.g. due to symptomatic gallstones, within the last 6 months, unless resolved following cholecystectomy
13. Inability to safely obtain a liver biopsy
14. Known human immunodeficiency virus (HIV) infection
15. Weight loss ≥ 10% within 6 months of Day 1
16. Use of controlled substances (including inhaled or injected drugs) or non-prescribed use of prescription drugs within 1 year of screening to the point of interfering with the subject's ability to comply with study procedures and study drug administration in the investigator's judgement
17. History of or active malignancies, other than those successfully treated with curative intent and believed to be cured
18. Significant systemic or major illness other than liver disease that in the opinion of the investigator would preclude the subject from participating in and completing the study, including but not limited to acute coronary syndrome or stroke within 6 months of screening or major surgery within 3 months of screening
19. History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QTcF interval >480 milliseconds (msec)
20. Prior or planned (during the time frame of the study) bariatric surgery
21. If female: planned or known pregnancy, positive urine or serum pregnancy test, or lactating/breastfeeding
22. Previous treatment with emricasan or active investigational medication in a clinical trial within 6 months prior to Day 1
23. Prior liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Fibrosis improvement by at least one stage without worsening of steatohepatitis | Week 72
  Proportion of subjects who improve fibrosis on liver biopsy by at least one stage without worsening of steatohepatitis in the emricasan group compared to placebo

SECONDARY OUTCOMES:
Steatohepatitis resolution (based on liver biopsy) | Baseline & Week 72
  The proportion of subjects who resolve steatohepatitis without worsening of fibrosis in the emricasan group compared to placebo
Improvement in the Non-alcoholic fatty liver disease (NAFLD) Activity Score | Baseline & Week 72
  The proportion of subjects who improve the NAFLD Activity Score (NAS), its components (steatosis, lobular inflammation, ballooning), and portal inflammation, in the emricasan group compared to placebo
Caspase 3/7 Relative Light Units and Alanine aminotransferase (ALT) | Day 1, week 4, 24, 48, and 72
  To asses whether emricasan compared to placebo improves biomarkers Caspase 3/7 RLU and ALT Unit/Liter (U/L) in subjects with NASH fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Chan, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (103):
- United States (83):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Clinical and Translational Sciences Research Center, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Fresno Clinical Research Center, Freestone, California
  - UCLA The Pfleger Liver Institute, Los Angeles, California
  - Gastrointestinal Biosciences, Los Angeles, California
  - Surinder Singh Saini, M.D., Inc., Newport Beach, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Florida Digestive Health Specialist, Lakewood Rch, Florida
  - Miami Veterans Administration Healthcare System, Miami, Florida
  - University of Miami/Schiff Center for Liver Diseases, Miami, Florida
  - Florida Hospital Orlando Transplant Institute, Orlando, Florida
  - Tampa General Medical Group, Tampa, Florida
  - iResearch Atlanta LLC, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Aquiant Research, New Albany, Indiana
  - Iowa Digestive Disease Center, P.C, Clive, Iowa
  - UnityPoint Clinic Center For Liver Disease, Des Moines, Iowa
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine-Infectious Disease Clinical Research Unit, St Louis, Missouri
  - Doctors Office Center, Newark, New Jersey
  - State University of New York, Buffalo, New York
  - Northwell Health, Inc., Manhasset, New York
  - Mount Sinai Beth Israel Medical Center, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center (CUMC), New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Carolinas Healthcare System, Center for Liver Disease, Charlotte, North Carolina
  - Duke University Medical Center, Duke South Clinics, Durham, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - PMG Research at Charleston, Charleston, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - Pinnacle Clinical Research, PLLC, Live Oak, Texas
  - American Research Corporation at the Texas Liver Institue, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Bon Secours Richmond Health System, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington
- Germany (9):
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bönning, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Eugastro GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Spain (11):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Goodman Z, Jabbar A, Vemulapalli R, Younes ZH, Freilich B, Sheikh MY, Schattenberg JM, Kayali Z, Zivony A, Sheikh A, Garcia-Samaniego J, Satapathy SK, Therapondos G, Mena E, Schuppan D, Robinson J, Chan JL, Hagerty DT, Sanyal AJ. A randomized, placebo-controlled trial of emricasan in patients with NASH and F1-F3 fibrosis. J Hepatol. 2020 May;72(5):816-827. doi: 10.1016/j.jhep.2019.11.024. Epub 2019 Dec 27. PMID 31887369